CLINICAL TRIAL: NCT06181760
Title: A Phase 1a, Randomized, Double-blind Placebo-controlled Study to Evaluate Safety and Tolerability and to Characterize the Pharmacokinetic Profile of Single Ascending Doses of Fenretinide Oral Capsules in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety of Fenretinide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Island Pharmaceuticals (Industry)
Collaborators: Beyond Drug Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISLA101-P01-CT001
Record Dates: First submitted 2023-10-25; First posted 2023-12-26 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Safety and Tolerability
MeSH Terms: interventions — Fenretinide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fenretinide 300 mg/m^2 (Active Comparator): Single oral dose of fenretinide, 300 mg/m^2 under fasted conditions (Phase 1)
  Interventions: Drug: Fenretinide
- Fenretinide 600 mg/m^2 (Active Comparator): Single oral dose of fenretinide, 600 mg/m^2 under fasted conditions (Phase 1)
  Once all groups finish Phase 1, return to complete Phase 2 with a single oral dose of fenretinide, 600 mg/m^2 under fed conditions per recommendation from the independent Safety Review Committee.
  Interventions: Drug: Fenretinide
- Fenretinide 900 mg/m^2 (Active Comparator): Single oral dose of fenretinide, 900 mg/m^2 under fasted conditions (Phase 1)
  Interventions: Drug: Fenretinide
- Placebo (Placebo Comparator): Single oral dose of placebo capsules under fasted conditions (Phase 1)
  Once all groups finish Phase 1, return to complete Phase 2 with a single oral dose of placebo capsules under fed conditions per recommendation from the independent Safety Review Committee.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenretinide — Ascending single doses of oral fenretinide
  Arms: Fenretinide 300 mg/m^2; Fenretinide 600 mg/m^2; Fenretinide 900 mg/m^2
Drug: Placebo — Single oral dose of matching placebo capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical trial was to learn about a single dose of fenretinide in healthy volunteers, in both a fasted and fed state. The main questions to answer were:

* How well is a single dose of fenretinide tolerated? AND
* How is a single dose of fenretinide metabolized in healthy volunteers?

Participants will be asked to:

* Remain confined in a clinical research unit for 5 days after dosing.
* Provide blood samples for intense PK sampling and safety labs.
* Fast for 10 hours prior to administration of study drug (fasted cohorts).
* Consume a high fat meal prior to administration of study drug (fed cohort).
* Return to the clinic for a single follow-up visit for safety assessments.

The study will compare active fenretinide to placebo to see if fenretinide is more or less tolerable than placebo.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled single ascending dose study. There are 3 planned dose-level cohorts (Cohorts 1-3). Each dose-level cohort will consist of 8 subjects (6 active + 2 placebo), who will be treated under fasted conditions. The subjects in the highest tolerated dose-level cohort (determined by the Safety Review Committee) will also be administered ISLA101 or placebo under fed conditions, in a cross-over manner (Cohort 4).

Proposed doses are 300, 600, and 900 mg/m^2 (equivalent to 8.1, 16.2, and 24.3 mg/kg). Each subject will be allocated to 1 dose level only.

The study will include a 5-day stay in the clinical research unit followed by a final safety follow-up visit at Day 8, where subjects will be under fasted conditions when they are dosed on Study Day 1.

For cohort 4, the study will again include a 5-day stay in the clinical research unit followed by a final safety follow-up visit at Day 17, where subjects will be under fed conditions when they are dosed on Study Day 10.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers not of childbearing potential, who are 18 years to 65 years of age (inclusive) at the time of signing the informed consent form (ICF).
2. Females not of childbearing potential, as defined in the following criteria:

   1. History of hysterectomy.
   2. Post-menopausal.

   i. Natural post-menopausal females with at least 12 months from natural spontaneous amenorrhea and a serum follicle-stimulating hormone (FSH) concentration ≥ 40 IU/L.

   ii. Post-surgical females must have undergone bilateral oophorectomy at least 6 weeks prior to study.
3. Male subjects with female partners of childbearing potential must agree to practice abstinence or use a combination of 2 of the following acceptable birth control methods during the study and for at least 90 days after dosing:

   1. Partners have an intrauterine device (IUD) without hormones in place for at least 3 months.
   2. Barrier method (condom or diaphragm) for at least 14 days prior to screening and 90 days after dosing with study drug.
   3. Partners using stable hormonal contraceptive for at least 3 months prior to screening and for 90 days after dosing with study drug.
   4. History of vasectomy at least 3 months prior to signing the ICF.
4. Must be able to understand and provide signed informed consent for study participation.
5. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
6. Body mass index (BMI) 18.0 to 32.0 kg/m2 (inclusive), and a body weight ≥ 50 kg.
7. Normal renal function, defined as estimated glomerular filtration rate (eGFR) ≥ 70 mL/min/1.73 m2 at screening and Day -1.
8. Clinical laboratory values should be within the laboratory's stated normal range. If not within this range, they must be without clinical significance, as determined by the Investigator.
9. No history of clinically relevant medical disorders, as determined by the Investigator.

Exclusion Criteria:

1. Known or suspected pregnancy (confirmed via a positive serum human chorionic gonadotropin [hCG] pregnancy test at screening), planned pregnancy during the study period, nursing, or lactation.
2. Women of childbearing potential or men who intend to father a child or donate sperm during the study period and for 3 months after study drug administration.
3. Known allergy to fenretinide or any of the components of ISLA101.
4. Evidence or history of clinically significant medical conditions, such as hematological, renal, endocrine (e.g., polycystic ovarian syndrome or other anovulatory states), immunologic, pulmonary, metabolic, gastrointestinal (e.g., Crohn's disease, acute or chronic pancreatitis, and others) and surgery (except for simple appendectomy or repair of a hernia), which all can influence the absorption of study drug; cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), or any other illness that the Investigator considers exclusionary or that could interfere with the interpretation of the study results.
5. History of severe infectious disease or recurrent infections.
6. Aspartate transaminase (AST), alanine aminotransferase (ALT), or total bilirubin above the 1.5 x upper limit of normal (ULN) at screening and Day -1.
7. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities at screening and Day -1, long QT syndrome, or a history of cardiac disease.
8. Abnormal diet that may affect absorption, distribution, metabolism, or excretion of drugs, for example, lacking standard nutrients (e.g, cleansing diet 2 weeks before or during the study).
9. Positive result for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening.
10. History of positive test for tuberculosis (TB) at screening.
11. A subject who has donated 1 unit of blood of over 500 mL within 56 days prior to the study drug administration, or donated plasma within 14 days prior to study drug administration.
12. Use of systemic antibiotics within 30 days prior to dosing.
13. Any use of drugs that inhibit or induce CYP enzymes within 30 days prior to administration of study drug and for the duration of study participation.
14. Use of any tobacco products, e-cigarettes, and/or nicotine replacement products in the 3 months preceding screening.
15. Any food allergy, intolerance, or restriction that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
16. Recent history of (within the past 12 months), or strong potential for, alcohol or substance abuse. Alcohol abuse will be defined as > 14 drinks per week (1 drink = 10g of ethanol).
17. History of drug or alcohol abuse within 5 years before screening or positive result of UDS (e.g, amphetamines, benzodiazepines, cannabinoids, cocaine, hallucinogens, opiates) or alcohol breath test at screening.
18. Exposure to any investigational agent or used an invasive investigational medical device within 30 days or within a period less than 5 drug half-lives prior to study entry (whichever is longer).
19. Study site employees, Sponsor's employees, or immediate family members of a study site or Sponsor employee.
20. Previously enrolled in this study.
21. Vaccination 14 days from screening or plans to get a vaccine within 30 days after dosing.
22. Acute infection (such as influenza) or relevant lesion at the time of Screening or Day -1. Subjects can be rescreened once they have recovered.
23. Criteria at the discretion of the Investigator:

    1. Chronic medical condition that impacts subject safety.
    2. Clinically significant abnormal physical examination or vital signs at screening.
    3. Condition believed to interfere with the subject's ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk.
    4. History or evidence of a clinically significant disorder, condition, or disease that that is believed to significantly impair pain perception (e.g., history of stroke, history of neuropathy), would pose a risk to subject safety or interfere with evaluation, procedures, or study completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Argent, MD, Principal Investigator — Scientia Clinical Research
Locations (1):
- Island Site 01, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 total subjects were enrolled in the study. After all fasted cohorts completed (i.e., 300 mg/m^2, 600 mg/m^2, 900 mg/m^2 as well as placebo) data was reviewed by the independent Safety Review Committee. The recommendation was to bring back the 600 mg/m^2 group to complete the fed cohort were only 4 out of the 6 subjects were available.
  Overall 25 subjects were enrolled, but there were 4 subjects (3 subjects on ISLA101 and 1 subject on placebo) that also participated in the fed cohort.
Groups:
- Fenretinide 300 mg/m^2: Single oral dose of fenretinide, 300 mg/m^2 under fasted conditions only
- Fenretinide 600 mg/m^2: Single oral dose of fenretinide, 600 mg/m^2 under fasted.
  Subjects completed a wash out period of at least 3 days.
  Subjects returned and took a Single oral dose of fenretinide, 600 mg/m^2 and fed conditions
- Fenretinide 900 mg/m^2: Single oral dose of fenretinide, 900 mg/m^2 under fasted conditions only
- Placebo: Single oral dose of placebo capsules
  Placebo: Single oral dose of matching placebo capsules under fasted conditions
  Subjects completed a washout period of at least 3 days.
  Subjects returned to complete the second intervention period taking a single oral dose of matching placebo capsules under fed conditions
Period: First Intervention (Fasted)
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo
Started | 6 | 6 | 6 | 7
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Second Intervention (Fed)
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo
Started | 0 | 3 | 0 | 1
Completed | 0 | 3 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 25 total subjects were enrolled in the study. After all fasted cohorts completed (i.e., 300 mg/m^2, 600 mg/m^2, 900 mg/m^2 as well as placebo) data was reviewed by the independent Safety Review Committee. The recommendation was to bring back the 600 mg/m^2 group to complete the fed cohort and only 4 out of the 6 subjects were available (i.e., 3 subjects on ISLA101 and 1 subject on placebo).
Groups:
- Fenretinide 600 mg/m^2: Single oral dose of fenretinide, 600 mg/m^2 under fasted and fed conditions
- Placebo: Single oral dose of placebo capsules under fasted and fed conditions
- Total: Total of all reporting groups
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.57 (10.443) | 40.23 (9.438) | 34.33 (13.049) | 30.66 (10.588) | 34.3 (10.872)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 2
  Male | 5 | 5 | 6 | 7 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 3 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 1 | 3 | 4 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 6 | 6 | 7 | 25
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.9 (4.35) | 26.3 (4.40) | 22.78 (2.79) | 24.31 (3.12) | 24.56 (3.69)

OUTCOME MEASURES:

1. Primary Outcome: Number and % of Subjects Experiencing Adverse Events Following a Single Oral Dose of Fenretinide Under Fasted Conditions
Time Frame: First Intervention (Day 1 to Day 8)
Population: 25 total subjects were enrolled in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Fenretinide 300 mg/m^2: Single oral dose of fenretinide, 300 mg/m^2 under fasted conditions
- Fenretinide 600 mg/m^2: Single oral dose of fenretinide, 600 mg/m^2 under fasted conditions
- Fenretinide 900 mg/m^2: Single oral dose of fenretinide, 900 mg/m^2 under fasted conditions
- Placebo: Single oral dose of placebo capsules under fasted conditions
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7
Participants | 1 | 2 | 3 | 2

2. Primary Outcome: Number and % of Subjects Experiencing Serious Adverse Events Following a Single Oral Dose of Fenretinide Under Fasted Conditions
Description: 25 total subjects were enrolled in the study.
Time Frame: First Intervention (Day 1 to Day 8)
Population: 25 total subjects were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Assess the CMax - Observed Maximum Plasma Concentration Following a Single Oral Dose of Fenretinide
Description: Secondary objective
Time Frame: First Intervention (Day 1 to Day 8), washout period, Second Intervention (Day 9-17)
Population: The PK Population was comprised of all subjects in the safety population who have a pre-dose PK sample and at least one post-dose analyzable PK sample and at least 1 post-dose analyzable PK sample (quantifiable Plasma concentration). Subjects in the placebo group did not have Cmax analyzed as they did not receive study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo: Single oral dose of placebo capsules
  Placebo: Single oral dose of matching placebo capsules
- Fenretinide 600 mg/m^2 (Fed): Single oral dose of fenretinide, 600 mg/m^2 under fed conditions
  Study Days 9-17
- Placebo (Fed): single oral doses of placebo under fed conditions
  Study Days 9-17
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo | Fenretinide 600 mg/m^2 (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 3 | 0
ng/mL | 195.8 (92.35) | 524.8 (74.2) | 624.2 (142.2) |  | 1455 (521.6) |

4. Secondary Outcome: Assess the TMax - Time to Reach Maximum Concentration Curve Following a Single Oral Dose of Fenretinide in the Fasted and Fed State
Description: 25 total subjects were enrolled in the study. After all fasted cohorts completed (i.e., 300 mg/m^2, 600 mg/m^2, 900 mg/m^2 as well as placebo) data was reviewed by the independent Safety Review Committee. The recommendation was to bring back the 600 mg/m^2 group to complete the fed cohort and only 4 out of the 6 subjects were available (i.e., 3 subjects on ISLA101 and 1 subject on placebo).
Time Frame: First Intervention (Day 1 to Day 8), washout period, Second Intervention (Day 9-17)
Population: The PK Population was comprised of all subjects in the safety population who have a pre-dose PK sample and at least one post-dose analyzable PK sample and at least 1 post-dose analyzable PK sample (quantifiable Plasma concentration). Subjects in the placebo group did not have Tmax analyzed as they did not receive study drug.
Measure: Mean (Full Range); unit: hours
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo | Fenretinide 600 mg/m^2 (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 3 | 0
hours | 5.895 [2.97 to 6.0] | 5.15 [5.07 to 6.02] | 5.015 [4.88 to 6.0] |  | 5.98 [5.98 to 9.97] |

5. Secondary Outcome: Assess the AUC-∞ Area Under the Concentration Curve From Zero to Infinite Time Following a Single Oral Dose of Fenretinide in the Fasted and Fed State
Description: as for outcome 4
Time Frame: First Intervention (Day 1 to Day 8), washout period, Second Intervention (Day 9-17)
Population: The PK Population was comprised of all subjects in the safety population who have a pre-dose PK sample and at least one post-dose analyzable PK sample and at least 1 post-dose analyzable PK sample (quantifiable Plasma concentration). Subjects in the placebo group did not have AUC-∞ analyzed as they did not receive study drug.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo | Fenretinide 600 mg/m^2 (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 3 | 0
h*ng/mL | 3479 (1947) | 8209 (836.9) | 9621 (2145) |  | 25800 (8726) |

6. Secondary Outcome: Assess the AUC(Last) - Area Under the Curve up to the Last Quantifiable Timepoint After a Single Oral Dose of Fenretinide in the Fasted and Fed State
Description: as for outcome 4
Time Frame: First Intervention (Day 1 to Day 8), washout period, Second Intervention (Day 9-17)
Population: The PK Population was comprised of all subjects in the safety population who have a pre-dose PK sample and at least one post-dose analyzable PK sample and at least 1 post-dose analyzable PK sample (quantifiable Plasma concentration). Subjects in the placebo group did not have AUC(last) analyzed as they did not receive study drug.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo | Fenretinide 600 mg/m^2 (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 3 | 0
h*ng/mL | 3212 (1795) | 7894 (844.6) | 9089 (2039) |  | 24460 (8395) |

7. Secondary Outcome: Assess the Half Life of a Single Oral Dose of Fenretinide in the Fasted and Fed State
Description: as for outcome 4
Time Frame: First Intervention (Day 1 to Day 8), washout period, Second Intervention (Day 9-17)
Population: The PK Population was comprised of all subjects in the safety population who have a pre-dose PK sample and at least one post-dose analyzable PK sample and at least 1 post-dose analyzable PK sample (quantifiable Plasma concentration). Subjects in the placebo group did not have half-life analyzed as they did not receive study drug.
Measure: Mean (Full Range); unit: hours
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo | Fenretinide 600 mg/m^2 (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 3 | 0
hours | 22.41 [9.788 to 35.73] | 28.21 [22.21 to 42.64] | 26.67 [21.23 to 29.47] |  | 27.77 [26.41 to 29.23] |

8. Primary Outcome: Number and % of Subjects Experiencing Adverse Events Following a Single Oral Dose of Fenretinide Under Fed Conditions
Description: Subjects in the 600 mg/m^2 came back to complete the fed cohort, as this was the only group to return based on the recommendations by the Safety Review Committee. Only 4 out of the 6 subjects returned for this cohort (i.e., 3 subjects on ISLA101 and 1 subject on placebo).
Time Frame: Second Intervention (Day 9 to Day 17)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Fenretinide 300 mg/m^2: Single oral dose of fenretinide, 300 mg/m^2 under fed conditions
- Fenretinide 600 mg/m^2: Single oral dose of fenretinide, 600 mg/m^2 under fed conditions
- Fenretinide 900 mg/m^2: Single oral dose of fenretinide, 900 mg/m^2 under fed conditions
- Placebo: Single oral dose of placebo capsules under fed conditions
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 1
Participants | 0 | 0 | 0 | 0

9. Primary Outcome: Number and % of Subjects Experiencing Serious Adverse Events Following a Single Oral Dose of Fenretinide Under Fed Conditions
Description: as for outcome 4
Time Frame: Second Intervention (Day 9 to 17)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Fenretinide 300 mg/m^2: Single oral dose of fenretinide, 300 mg/m^2 under fed conditions only
- Fenretinide 900 mg/m^2: Single oral dose of fenretinide, 900 mg/m^2 under fed conditions only
Arm/Group | Fenretinide 300 mg/m^2 | Fenretinide 600 mg/m^2 | Fenretinide 900 mg/m^2 | Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 1
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored throughout the study for adverse reactions to the study drug and/or procedures from the time of informed consent through end of study (either through Day 8 for the fasted cohorts or through Day 17 for the fed cohort).
Groups:
- Fenretinide 300 mg/m^2 (First Intervention): Single oral dose of fenretinide, 300 mg/m^2 under fasted conditions
- Fenretinide 600 mg/m^2 (First Intervention): Single oral dose of fenretinide, 600 mg/m^2 under fasted conditions
- Fenretinide 900 mg/m^2 (First Intervention): Single oral dose of fenretinide, 900 mg/m^2 under fasted conditions
- Placebo (First Intervention): Single oral dose of placebo capsules under fasted conditions
- Fenretinide 600 mg/m^2 (Second Intervention): Single oral dose of fenretinide, 600 mg/m^2 under fed conditions
- Placebo (Second Intervention): Single oral dose of placebo capsules under fed conditions
Arm/Group | Fenretinide 300 mg/m^2 (First Intervention) | Fenretinide 600 mg/m^2 (First Intervention) | Fenretinide 900 mg/m^2 (First Intervention) | Placebo (First Intervention) | Fenretinide 600 mg/m^2 (Second Intervention) | Placebo (Second Intervention)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/6 | 2/7 | 0/3 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenretinide 300 mg/m^2 (First Intervention) (N=6) | Fenretinide 600 mg/m^2 (First Intervention) (N=6) | Fenretinide 900 mg/m^2 (First Intervention) (N=6) | Placebo (First Intervention) (N=7) | Fenretinide 600 mg/m^2 (Second Intervention) (N=3) | Placebo (Second Intervention) (N=1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vascular access site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma muscle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT06181760/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT06181760/SAP_001.pdf